CLINICAL TRIAL: NCT02673736
Title: A Phase 1 Study to Assess Safety, Pharmacokinetics, and Pharmacodynamics of PLX73086 as a Single Agent in Subjects With Advanced Solid Tumors and in Subjects With Locally Advanced or Refractory Tenosynovial Giant Cell Tumor (TGCT)
Brief Title: A Study of PLX73086 in Advanced Solid Tumors and Locally Advanced or Refractory Tenosynovial Giant Cell Tumor
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Discontinued
Sponsor: Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX123-01
Record Dates: First submitted 2016-01-29; First posted 2016-02-04 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Solid Tumors; Tenosynovial Giant Cell Tumor; Synovitis, Pigmented Villonodular
Keywords: PLX73086; Synovitis, Pigmented Villonodular; Tenosynovial Giant Cell Tumor; Joint Diseases; Neoplasms; Synovitis
MeSH Terms: conditions — Giant Cell Tumor of Tendon Sheath; Synovitis, Pigmented Villonodular; Joint Diseases; Neoplasms; Synovitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PLX73086 (Experimental): Part 1: Open-label, sequential PLX73086 dose escalation in approximately 36 solid tumors subjects.
  Part 2: Extension cohort at the recommended phase 2 dose (RP2D) of PLX73086 in approximately 30 subjects with histologically confirmed, unresectable, locally advanced or refractory TGCT (including metastatic disease).
  Interventions: Drug: PLX73086

INTERVENTIONS:
Drug: PLX73086

SUMMARY:
The purpose of this research study is to evaluate safety, pharmacokinetics and preliminary efficacy of the investigational drug PLX73086 in subjects with solid tumors including subjects with locally advanced or refractory tenosynovial giant cell tumor (TGCT).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Part 1: Subjects with solid tumors that are refractory to, relapsed after or intolerant to standard therapy, or for whom no standard therapy exists or who are considered by the investigator to be inappropriate for standard therapy.
* Part 2: Subjects with histologically confirmed, locally advanced or refractory TGCT (including metastatic disease) that has been deemed unresectable by an orthopedic surgeon or similar qualified personnel.
* Measurable disease by RECIST 1.1 criteria.
* Women of child-bearing potential must have a negative pregnancy test within 7 days prior to initiation of dosing and must agree to use an acceptable method of birth control from the time of the negative pregnancy test up to 3 months after the last dose of study drug, Fertile men must also agree to use an acceptable method of birth control while on study drug and up to 3 months after the last dose of study drug.
* All associated toxicity from previous or concurrent cancer therapy must be resolved (to ≤ Grade 1 or Baseline) prior to study treatment administration.
* Willingness and ability to provide written informed consent prior to any study-related procedures and comply with all study requirements.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
* Life expectancy ≥ 3 months.
* Adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

* Symptomatic brain metastases.
* Investigational drug use within 14 days (or 5 half-lives, whichever is longer) of the first dose of PLX73086.
* Major surgical procedure, open biopsy (excluding skin cancer resection), or significant traumatic injury within 14 days of initiating study drug (unless the wound has healed) or anticipation of the need for major surgery during the study.
* Active secondary malignancy unless the malignancy is not expected to interfere with the evaluation of safety and is approved by the Medical Monitor. Examples of the latter include basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, and isolated elevation of prostate-specific antigen. Subjects with a completely treated prior malignancy and no evidence of disease for ≥ 2 years are eligible.
* Inability to take oral medication or significant nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption.
* Baseline mean QTcF ≥ 450 msec (for males) or ≥ 470 msec (for females) at Screening.
* Clinically significant cardiac arrhythmias including bradyarrhythmias and/or subjects who require anti-arrhythmic therapy (excluding beta blockers or digoxin). Subjects with controlled atrial fibrillation are not excluded
* Congenital long QT syndrome or subjects taking concomitant medications known to prolong the QT interval (e.g., tricyclics, azithromycin, methadone).
* History of clinically significant cardiac disease or congestive heart failure > New York Heart Association (NYHA) class 2. Subjects must not have unstable angina (anginal symptoms at rest) or new-onset angina within the last 3 months or myocardial infarction within the past 6 months.
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months before start of study medication (except for adequately treated catheter-related venous thrombosis occurring more than 1 month before the start of study medication).
* Strong CYP3A4 inhibitors or inducers as well as inhibitors of breast cancer resistance protein (BCRP) within 14 days or 5 drug half-lives, whichever is longer, before start of study drug.
* Subjects with > Grade 1 (high or low) serum potassium, magnesium, or calcium levels.
* Women who are breast-feeding or pregnant.
* Non-healing wound, ulcer, or bone fracture.
* Known HIV-positive individuals on combination antiretroviral therapy.
* Subjects with known active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy.
* Uncontrolled intercurrent illness (i.e., active infection ≥ Grade 2) or concurrent condition that, in the opinion of the Investigator, would interfere with the study endpoints or the subject's ability to participate.
* The presence of a medical or psychiatric condition that, in the opinion of the Principal Investigator, makes the subject inappropriate for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-02; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Safety of PLX73086, as measured by adverse events and serious adverse events [Part 1 and Part 2 of research study] | 1 year
Area under the concentration-time curve (AUC) of PLX73086 [Part 1 of research study] | 1 year
Maximum observed concentration (Cmax) of PLX73086 [Part 1 of research study] | 1 year
Time to peak concentration (Tmax) of PLX73086 [Part 1 of research study] | 1 year
Half life (t1/2) of PLX73086 [Part 1 of research study] | 1 year

SECONDARY OUTCOMES:
Efficacy of PLX73086 measured by overall response rate (ORR) [Part 1 of research study] | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - HonorHealth, Scottsdale, Arizona
  - Karmanos Cancer Institute, Detroit, Michigan
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided